CLINICAL TRIAL: NCT07367191
Title: The Role of Temporal Changes in Pain Response After Transforaminal Epidural Steroid Injection on Treatment Success
Status: Not yet recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MarmaraU-FTR-OK-3
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Lumbar Disc Herniation; Lumbar Radiculopathy; Radicular Low Back Pain; Sciatica
Keywords: TFESI; Temporal Pain Response; Numeric Rating Scale; NRS; Transforaminal Epidural Steroid Injection; Treatment Success
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy; Sciatica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Receiving Treatment for Lumbar Disc Herniation-Related Radiculopathy: Adult patients with lumbar disc herniation-related radiculopathy undergoing routine fluoroscopy-guided transforaminal epidural steroid injection as part of standard clinical care, followed prospectively for pain outcomes.
  Interventions: Procedure: Transforaminal epidural steroid injection

INTERVENTIONS:
Procedure: Transforaminal epidural steroid injection — Fluoroscopy-guided transforaminal epidural steroid injection performed as part of routine clinical care. After confirmation of correct needle placement with contrast medium and exclusion of intravascular uptake, a mixture of betamethasone, bupivacaine, and normal saline is injected slowly into the epidural space. This procedure is not assigned by the study and is performed according to standard clinical practice.

SUMMARY:
Transforaminal epidural steroid injection (TFESI) is a commonly used minimally invasive procedure for the treatment of lumbar radicular pain secondary to disc herniation. Although TFESI has been shown to provide significant pain relief in a substantial proportion of patients, the onset, duration, and temporal pattern of pain relief after the procedure vary considerably among individuals. The relationship between early pain response patterns and long-term treatment success remains poorly understood.

This prospective observational study aims to evaluate whether temporal changes in pain intensity following TFESI, particularly during the early post-procedural period, are associated with clinical treatment success at mid- and long-term follow-up. Pain intensity will be assessed using the Numeric Rating Scale (NRS) at predefined time points following the procedure, and treatment success will be defined as a ≥50% reduction in NRS score compared with baseline.

DETAILED DESCRIPTION:
Transforaminal epidural steroid injection (TFESI) is widely utilized in patients with lumbar disc herniation-related radiculopathy who do not respond adequately to conservative treatment and are not immediate candidates for surgery. While previous studies have demonstrated the overall effectiveness of TFESI, there is limited evidence regarding the temporal characteristics of pain relief following the procedure and how these patterns influence long-term outcomes.

In routine clinical practice, patients may exhibit heterogeneous pain trajectories after TFESI, including early responders, delayed responders, transient responders, or those with minimal or no response. Identifying early pain response patterns that predict treatment success may help clinicians optimize patient counseling, follow-up strategies, and decisions regarding repeat interventions.

In this prospective observational cohort study, adult patients undergoing fluoroscopy-guided TFESI as part of routine clinical care will be followed longitudinally. Pain intensity will be assessed using the Numeric Rating Scale (NRS) before the procedure; at 1 hour post-procedure; every 72 hours during the first 21 days; and at 1, 3, and 6 months. Demographic data, clinical characteristics, and radiological findings from lumbar magnetic resonance imaging will be recorded.

The primary objective is to determine whether early temporal changes in pain intensity following TFESI are associated with treatment success at 3 months. Secondary objectives include evaluating treatment success at 6 months and identifying early pain response thresholds that predict favorable outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Pre-procedural Numeric Rating Scale (NRS) pain score of 4 or higher
* Presence of segmental lumbar disc herniation demonstrated on magnetic resonance imaging (MRI) consistent with clinical findings
* Undergoing fluoroscopy-guided transforaminal epidural steroid injection due to insufficient response to conservative treatments, as determined by the algology clinic

Exclusion Criteria:

* Presence of spondylolisthesis, scoliosis, or lumbar spinal stenosis accompanying lumbar disc herniation
* Presence of malignancy
* History of lumbar spine surgery for disc herniation
* Transforaminal epidural steroid injection within the previous 6 months
* Requirement for repeat epidural steroid injection during the data collection or follow-up period
* Inability to be contacted for follow-up assessments by telephone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 to 65 years with lumbar disc herniation-related radiculopathy who are undergoing fluoroscopy-guided transforaminal epidural steroid injection as part of routine clinical care. All participants have clinically significant radicular pain with a pre-procedural Numeric Rating Scale (NRS) score of 4 or higher and lumbar disc herniation confirmed by magnetic resonance imaging (MRI) at a segmental level consistent with clinical findings.
  Patients included in the study are those who have not achieved adequate symptom relief with conservative treatment modalities and are therefore referred for transforaminal epidural steroid injection by the algology clinic. Participants are prospectively followed after the procedure to evaluate temporal changes in pain intensity and their association with clinical treatment success.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-08-16 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Role of Early Temporal Changes in Pain Response on Treatment Success | Baseline to 6 months after transforaminal epidural steroid injection
  Association between temporal changes in pain response following transforaminal epidural steroid injection and clinical treatment success.
  Pain intensity will be assessed using the Numeric Rating Scale (NRS) at baseline (pre-procedure), at 1 hour post-procedure via face-to-face assessment, every 72 hours during the first 21 days, and at 1, 3, and 6 months via telephone follow-up. Temporal patterns of pain response over these time points will be analyzed in relation to clinical treatment success, defined as a ≥50% reduction in NRS score at 3 months compared with baseline.Clinical treatment success is defined as a ≥50% reduction in NRS score at 3 months compared with baseline.

SECONDARY OUTCOMES:
Clinical Treatment Success at 3 Months | 3 months after transforaminal epidural steroid injection
  Proportion of participants achieving a ≥50% reduction in Numeric Rating Scale (NRS) pain score at 3 months compared with baseline (pre-procedure).
Clinical Treatment Success at 6 Months | 6 months after transforaminal epidural steroid injection
  Proportion of participants achieving a ≥50% reduction in Numeric Rating Scale (NRS) pain score at 6 months compared with baseline.
Time to Maximum Pain Relief | Up to 6 months after the procedure
  Time (in days) from transforaminal epidural steroid injection to the lowest recorded Numeric Rating Scale (NRS) pain score during follow-up.
Association Between Radiological Findings and Pain Response | Baseline to 6 months
  Relationship between lumbar magnetic resonance imaging characteristics (disc herniation level, location, size, and nerve root compression) and temporal pain response patterns following transforaminal epidural steroid injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara Üniversitesi Tıp Fakültesi, Istanbul, Maltepe 34854, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No